CLINICAL TRIAL: NCT01252563
Title: NORVASC10MG DRUG USE INVESTIGATION
Brief Title: Amlodipine 10mg Drug Use Investigation
Acronym: ENTER10
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0531097
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: ENTER10; Hypertension; Japanese; Norvasc 10mg; Post Marketing surveillance
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Amlodipine 10mg Tablet: Subjects taking Amlodipine 10mg Tablet.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Usual adult dosage is 2.5-5 mg of amlodipine given orally as a single daily dose. Dosage should be adjusted depending on the patient's symptoms. The dose can be raised up to 10 mg once daily for patients who show inadequate response.
  Other Names: Norvasc

SUMMARY:
In this survey, to collect the safety and efficacy information in the subjects who have been treated with amlodipine 5mg at least 4 weeks in daily practice.

DETAILED DESCRIPTION:
All the subjects whom an investigator prescribes Amlodipine (Norvasc®) 10mg Tablet should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who have been treated with amlodipine 5mg at least 4 weeks
* The subjects who had not achieved target BP

Exclusion Criteria:

* Subjects who have been prescribed amlodipine (Norvasc®) 10mg Tablet before

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects who have been treated with amlodipine 5mg at least 4 weeks and had not achieved target BP.
Sampling Method: Probability Sample
Enrollment: 14141 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531097&StudyName=Amlodipine%2010mg%20Drug%20Use%20Investigation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14141 participants were registered in the study. Of the 14141 participants, 366 participants were excluded from the study because their case report forms were not collected, mainly due to the lack of cooperation from the investigators. Finally, 13775 participants were included in the study.
Groups:
- Amlodipine 10 mg Tablet: Participants taking Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Amlodipine 10 mg Tablet
Started | 13775
Completed | 13343
Not Completed | 432
Not completed — Contract Deviation | 41
Not completed — Centralized Registration Deviation | 30
Not completed — Lost to Follow-up | 161
Not completed — No visit after first day of treatment | 194
Not completed — No drug administration | 6

BASELINE CHARACTERISTICS:
Population: A total of 13775 participants completed the survey. Of the 13775 participants, a total of 432 participants were excluded from the baseline analysis for the following reasons: no visit after first day of treatment, lost to follow up, contract deviation, centralized registration deviation and no drug administration.
Arm/Group | Amlodipine 10 mg Tablet
Number analyzed (Participants) | 13343
Age, Customized [Number; unit: Participants]
  <65 years | 5229
  >=65 years | 8114
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5839
  Male | 7504

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Amlodipine Tablets or Amlodipine OD Tablets at 10 mg/day. Relatedness to Amlodipine Tablets or Amlodipine OD Tablets was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: The safety analysis population comprised participants who had taken Amlodipine Tablets or Amlodipine OD Tablets at 10 mg/day at least once after the start of treatment.
Measure: Number; unit: participants
Arm/Group | Amlodipine 10 mg Tablet
Number analyzed (Participants) | 13343
participants | 208

2. Primary Outcome: The Achievement Rate to Ambulatory Blood Pressure Goal
Description: The achievement rates to ambulatory blood pressure goal specified in the Japanese guidelines (JSH2009) were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: The efficacy analysis population consisted of the participants, among the safety analysis population, who had their SBP/DBP measurement prior to the start of treatment and at least one post-baseline SBP/DBP measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- The Achievement Rate to Ambulatory Blood Pressure Goal: The achievement rates to ambulatory blood pressure goal specified in the Japanese guidelines (JSH2009) were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | The Achievement Rate to Ambulatory Blood Pressure Goal
Number analyzed (Participants) | 13124
Percentage of participants
  Week 4: number analyzed (Participants) | 9655
  Week 4 | 35.1 [34.2 to 36.1]
  Week 8: number analyzed (Participants) | 9534
  Week 8 | 40.1 [39.1 to 41.0]
  Week 12: number analyzed (Participants) | 8958
  Week 12 | 43.9 [42.8 to 44.9]
  Last Day: number analyzed (Participants) | 12987
  Last Day | 43.9 [43.0 to 44.7]

3. Primary Outcome: Changes in Ambulatory Systolic Blood Pressure From Baseline
Description: Changes in ambulatory systolic blood pressure (SBP) from baseline were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Changes in Ambulatory SBP From Baseline: changes in ambulatory SBP from baseline at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | Changes in Ambulatory SBP From Baseline
Number analyzed (Participants) | 13124
mmHg
  Week 4: number analyzed (Participants) | 9637
  Week 4 | -16.8 (15.20)
  Week 8: number analyzed (Participants) | 9520
  Week 8 | -18.4 (15.90)
  Week 12: number analyzed (Participants) | 8948
  Week 12 | -19.9 (16.05)
  Last Day: number analyzed (Participants) | 12963
  Last Day | -20.1 (16.31)
Statistical Analysis 1: Comparison: Changes in Ambulatory SBP From Baseline; The null hypothesis was that the mean change in ambulatory SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 4; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: Changes in Ambulatory SBP From Baseline; The null hypothesis was that the mean change in ambulatory SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 8; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: Changes in Ambulatory SBP From Baseline; The null hypothesis was that the mean change in ambulatory SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 12; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: Changes in Ambulatory SBP From Baseline; The null hypothesis was that the mean change in ambulatory SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Last Day; A one-sided paired t-test was performed to test the hypothesis

4. Primary Outcome: Changes in Ambulatory Diastolic Blood Pressure From Baseline
Description: Changes in ambulatory diastolic blood pressure (DBP) from baseline were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Changes in Ambulatory DBP From Baseline: changes in ambulatory DBP from baseline at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | Changes in Ambulatory DBP From Baseline
Number analyzed (Participants) | 13124
mmHg
  Week 4: number analyzed (Participants) | 9633
  Week 4 | -8.2 (10.47)
  Week 8: number analyzed (Participants) | 9514
  Week 8 | -9.1 (10.75)
  Week 12: number analyzed (Participants) | 8944
  Week 12 | -9.9 (11.03)
  Last Day: number analyzed (Participants) | 12958
  Last Day | -10.0 (11.06)
Statistical Analysis 1: Comparison: Changes in Ambulatory DBP From Baseline; The null hypothesis was that the mean change in ambulatory DBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 4; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: Changes in Ambulatory DBP From Baseline; The null hypothesis was that the mean change in ambulatory DBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 8; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: Changes in Ambulatory DBP From Baseline; The null hypothesis was that the mean change in ambulatory DBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 12; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: Changes in Ambulatory DBP From Baseline; The null hypothesis was that the mean change in ambulatory DBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Last Day; A one-sided paired t-test was performed to test the hypothesis

5. Secondary Outcome: Number of Participants With Adverse Events Listed in Japanese Package Insert
Description: Adverse events refer to all events undesirable for participants that occur after the start of treatment with Amlodipine Tablets or Amlodipine OD Tablets at 10 mg/day, regardless of presence/absence of causal relationship with Amlodipine Tablets or Amlodipine OD Tablets (including clinically significant abnormal changes in laboratory test values).
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Amlodipine 10 mg Tablet
Number analyzed (Participants) | 13343
participants | 566

6. Secondary Outcome: Number of Treatment Related Adverse Events Unlisted in Japanese Package Insert
Description: as for outcome 1
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Amlodipine 10 mg Tablet
Number analyzed (Participants) | 13343
Events | 21

7. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: With/Without Complication(s)
Description: To determine whether having complication(s) was a significant risk factor likely to affect the frequency of treatment-related adverse events. Complications included dyslipidemia, diabetes mellitus, metabolic syndrome, chronic kidney disease, angina pectoris, cerebrovascular disease, and myocardial infarction.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Complication(s): Participants who had at least one complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Without Complication(s): Participants who had no complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | With Complication(s) | Without Complication(s)
Number analyzed (Participants) | 9177 | 4166
Participants | 170 | 38
Statistical Analysis 1: Comparison: With Complication(s) vs Without Complication(s); The risk factor tested was "Complication". The null hypothesis was that there was no difference between participants with complication(s) and participants without complication in the frequency of treatment-related adverse events; Test type: Superiority or Other; p < 0.001, Chi-squared

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: Male vs. Female
Description: To determine whether gender was a significant risk factor likely to affect the frequency of treatment-related adverse events.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Male: Male participants who experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Female: Female participants who experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | Male | Female
Number analyzed (Participants) | 7504 | 5839
Participants | 87 | 121
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis was that there was no difference between male and female in the frequency of treatment-related adverse events; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: With/Without Complication (Angina Pectoris)
Description: To determine whether having angina pectoris as a complication was a significant risk factor likely to affect the frequency of treatment-related adverse events.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Angina Pectoris: Participants who had angina pectoris as a complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Without Angina Pectoris: Participants who had no angina pectoris as a complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | With Angina Pectoris | Without Angina Pectoris
Number analyzed (Participants) | 872 | 12471
Participants | 21 | 187
Statistical Analysis 1: Comparison: With Angina Pectoris vs Without Angina Pectoris; The risk factor tested was "angina pectoris" as a complication. The null hypothesis was that there was no difference between participants with angina pectoris and participants without angina pectoris in the frequency of treatment-related adverse events; Test type: Superiority or Other; p = 0.036, Chi-squared

10. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: With/Without Complication (Dyslipidaemia)
Description: To determine whether having dyslipidaemia as a complication was a significant risk factor likely to affect the frequency of treatment-related adverse events.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Dyslipidaemia: Participants who had dyslipidaemia as a complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Without Dyslipidaemia: Participants who had no dyslipidaemia as a complication and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | With Dyslipidaemia | Without Dyslipidaemia
Number analyzed (Participants) | 5308 | 8035
Participants | 99 | 109
Statistical Analysis 1: Comparison: With Dyslipidaemia vs Without Dyslipidaemia; The risk factor tested was "dyslipidaemia" as a complication. The null hypothesis was that there was no difference between participants with dyslipidaemia and participants without dyslipidaemia in the frequency of treatment-related adverse events; Test type: Superiority or Other; p = 0.020, Chi-squared

11. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: With/Without Concomitant Drug (Antihypertensive)
Description: To determine whether receiving antihypertensive as a concomitant drug was a significant risk factor likely to affect the frequency of treatment-related adverse events.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With Antihypertensive: Participants who received antihypertensive as a concomitant drug and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Without Antihypertensive: Participants who received no antihypertensive as a concomitant drug and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | With Antihypertensive | Without Antihypertensive
Number analyzed (Participants) | 7834 | 5509
Participants | 136 | 72
Statistical Analysis 1: Comparison: With Antihypertensive vs Without Antihypertensive; The risk factor tested was "antihypertensive" as a concomitant drug. The null hypothesis was that there was no difference between participants receiving antihypertensive and participants receiving no antihypertensive in the frequency of treatment-related adverse events; Test type: Superiority or Other; p = 0.049, Chi-squared

12. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events: With/Without Concomitant Drug (ARB)
Description: To determine whether receiving ARB as a concomitant drug was a significant risk factor likely to affect the frequency of treatment-related adverse events.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- With ARB: Participants who received ARB as a concomitant drug and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
- Without ARB: Participants who received no ARB as a concomitant drug and experienced treatment-related adverse events after having received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert at least once.
Arm/Group | With ARB | Without ARB
Number analyzed (Participants) | 6641 | 6702
Participants | 118 | 90
Statistical Analysis 1: Comparison: With ARB vs Without ARB; The risk factor tested was "ARB" as a concomitant drug. The null hypothesis was that there was no difference between participants receiving ARB and participants receiving no ARB in the frequency of treatment-related adverse events; Test type: Superiority or Other; p = 0.043, Chi-squared

13. Secondary Outcome: Number of Participants Who Achieved the Target Blood Pressure: With/Without Complication (Diabetes Mellitus)
Description: To determine whether having diabetes mellitus as a complication was a significant risk factor likely to affect the efficacy. The achievement rates to the target blood pressure specified in the Japanese guidelines (JSH2009) were calculated on the last day of the observation period.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- With Diabetes Mellitus: Participants with diabetes mellitus as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- Without Diabetes Mellitus: Participants without diabetes mellitus as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Arm/Group | With Diabetes Mellitus | Without Diabetes Mellitus
Number analyzed (Participants) | 2247 | 7004
Participants | 52 | 892
Statistical Analysis 1: Comparison: With Diabetes Mellitus vs Without Diabetes Mellitus; The risk factor tested was "diabetes mellitus" as a complication. The null hypothesis was that there was no difference between participants with diabetes mellitus and participants without diabetes mellitus in the efficacy; Test type: Superiority or Other; p < 0.001, Chi-squared

14. Secondary Outcome: Number of Participants Who Achieved the Target Blood Pressure: With/Without Complication (Chronic Kidney Disease)
Description: To determine whether having chronic kidney disease as a complication was a significant risk factor likely to affect the efficacy. The achievement rates to the target blood pressure specified in the Japanese guidelines (JSH2009) were calculated on the last day of the observation period.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- With Chronic Kidney Disease: Participants with chronic kidney disease as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- Without Chronic Kidney Disease: Participants without chronic kidney disease as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Arm/Group | With Chronic Kidney Disease | Without Chronic Kidney Disease
Number analyzed (Participants) | 1034 | 8217
Participants | 24 | 920
Statistical Analysis 1: Comparison: With Chronic Kidney Disease vs Without Chronic Kidney Disease; The risk factor tested was "chronic kidney disease" as a complication. The null hypothesis was that there was no difference between participants with chronic kidney disease and participants without chronic kidney disease in the efficacy; Test type: Superiority or Other; p < 0.001, Chi-squared

15. Secondary Outcome: Number of Participants Who Achieved the Target Blood Pressure: With/Without Complication (Myocardial Infarction)
Description: To determine whether having myocardial infarction as a complication was a significant risk factor likely to affect the efficacy. The achievement rates to the target blood pressure specified in the Japanese guidelines (JSH2009) were calculated on the last day of the observation period.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- With Myocardial Infarction: Participants with myocardial infarction as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- Without Myocardial Infarction: Participants without myocardial infarction as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Arm/Group | With Myocardial Infarction | Without Myocardial Infarction
Number analyzed (Participants) | 55 | 9196
Participants | 1 | 943
Statistical Analysis 1: Comparison: With Myocardial Infarction vs Without Myocardial Infarction; The risk factor tested was "myocardial infarction" as a complication. The null hypothesis was that there was no difference between participants with myocardial infarction and participants without myocardial infarction in the efficacy; Test type: Superiority or Other; p = 0.039, Chi-squared

16. Secondary Outcome: Number of Participants Who Achieved the Target Blood Pressure: With/Without Complication (Metabolic Syndrome)
Description: To determine whether having metabolic syndrome as a complication was a significant risk factor likely to affect the efficacy. The achievement rates to the target blood pressure specified in the Japanese guidelines (JSH2009) were calculated on the last day of the observation period.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- With Metabolic Syndrome: Participants with metabolic syndrome as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- Without Metabolic Syndrome: Participants without metabolic syndrome as a complication who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Arm/Group | With Metabolic Syndrome | Without Metabolic Syndrome
Number analyzed (Participants) | 1716 | 7535
Participants | 92 | 852
Statistical Analysis 1: Comparison: With Metabolic Syndrome vs Without Metabolic Syndrome; The risk factor tested was "metabolic syndrome" as a complication. The null hypothesis was that there was no difference between participants with metabolic syndrome and participants without metabolic syndrome in the efficacy; Test type: Superiority or Other; p < 0.001, Chi-squared

17. Secondary Outcome: Number of Participants Who Achieved the Target Blood Pressure: Ambulatory Systolic Blood Pressure
Description: To determine whether ambulatory systolic blood pressure at baseline was a significant risk factor likely to affect the efficacy. The achievement rates to the target blood pressure specified in the Japanese guidelines (JSH2009) were calculated on the last day of the observation period.
Time Frame: Last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- <120 mmHg at Baseline: Participants with ambulatory SBP of below 120 mmHg at baseline who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- 120 to 140 mmHg at Baseline: Participants with ambulatory SBP of 120 to 140 mmHg at baseline who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- 140 to 160 mmHg at Baseline: Participants with ambulatory SBP of 140 to 160 mmHg at baseline who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- 160 to 180 mmHg at Baseline: Participants with ambulatory SBP of 160 to 180 mmHg at baseline who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
- >= 180 mmHg at Baseline: Participants with ambulatory SBP of 180 mmHg or above at baseline who received Amlodipine Tablets or Amlodipine OD Tablets 10 mg/day orally according to Japanese Package Insert.
Arm/Group | <120 mmHg at Baseline | 120 to 140 mmHg at Baseline | 140 to 160 mmHg at Baseline | 160 to 180 mmHg at Baseline | >= 180 mmHg at Baseline
Number analyzed (Participants) | 82 | 863 | 4675 | 2808 | 757
Participants | 19 | 171 | 543 | 182 | 26
Statistical Analysis 1: Comparison: <120 mmHg at Baseline vs 120 to 140 mmHg at Baseline vs 140 to 160 mmHg at Baseline vs 160 to 180 mmHg at Baseline vs >= 180 mmHg at Baseline; The risk factor tested was "ambulatory SBP at baseline". The null hypothesis was that there was no association between ambulatory SBP at baseline and the number of participants who achieved the target blood pressure specified in the guidelines; Test type: Superiority or Other; p < 0.001, Chi-squared

18. Secondary Outcome: The Achievement Rate to Home Blood Pressure Goal
Description: The achievement rates to home blood pressure goal specified in the Japanese guidelines (JSH2009) were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- The Achievement Rate to Home Blood Pressure Goal: The achievement rates to home blood pressure goal specified in the Japanese guidelines (JSH2009) were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | The Achievement Rate to Home Blood Pressure Goal
Number analyzed (Participants) | 13124
Percentage of participants
  Week 4: number analyzed (Participants) | 2841
  Week 4 | 21.2 [19.7 to 22.8]
  Week 8: number analyzed (Participants) | 2675
  Week 8 | 27.9 [26.2 to 29.6]
  Week 12: number analyzed (Participants) | 2543
  Week 12 | 32.2 [30.4 to 34.1]
  Last Day: number analyzed (Participants) | 4265
  Last Day | 31.3 [29.9 to 32.7]

19. Secondary Outcome: Changes in Home Systolic Blood Pressure From Baseline
Description: Changes in home systolic blood pressure (SBP) from baseline were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Changes in Home SBP From Baseline: Mean changes in home SBP from baseline at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | Changes in Home SBP From Baseline
Number analyzed (Participants) | 13124
mmHg
  Week 4: number analyzed (Participants) | 2427
  Week 4 | -15.7 (13.34)
  Week 8: number analyzed (Participants) | 2302
  Week 8 | -18.0 (13.80)
  Week 12: number analyzed (Participants) | 2183
  Week 12 | -19.9 (14.38)
  Last Day: number analyzed (Participants) | 3494
  Last Day | -19.6 (14.27)
Statistical Analysis 1: Comparison: Changes in Home SBP From Baseline; The null hypothesis was that the mean change in home SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 4; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: Changes in Home SBP From Baseline; The null hypothesis was that the mean change in home SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 8; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: Changes in Home SBP From Baseline; The null hypothesis was that the mean change in home SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 12; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: Changes in Home SBP From Baseline; The null hypothesis was that the mean change in home SBP from the baseline was equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Last Day; A one-sided paired t-test was performed to test the hypothesis

20. Secondary Outcome: Changes in Home Diastolic Blood Pressure From Baseline
Description: Changes in home diastolic blood pressure (DBP) from baseline were calculated at weeks 4, 8, and 12 as well as on the last day of the observation period.
Time Frame: 4, 8, 12 weeks and last day of observation period (average of 14.76 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Changes in Home Diastolic Blood Pressure From Baseline: Mean changes in home DBP from baseline at weeks 4, 8, and 12 as well as on the last day of the observation period.
Arm/Group | Changes in Home Diastolic Blood Pressure From Baseline
Number analyzed (Participants) | 13124
mmHg
  Week 4: number analyzed (Participants) | 2332
  Week 4 | -8.3 (9.21)
  Week 8: number analyzed (Participants) | 2209
  Week 8 | -9.5 (9.46)
  Week 12: number analyzed (Participants) | 2126
  Week 12 | -10.4 (10.07)
  Last Day: number analyzed (Participants) | 3330
  Last Day | -10.4 (9.82)
Statistical Analysis 1: Comparison: Changes in Home Diastolic Blood Pressure From Baseline; The null hypothesis was that the mean changes in home DBP from the baseline are equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 4; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: Changes in Home Diastolic Blood Pressure From Baseline; The null hypothesis was that the mean changes in home DBP from the baseline are equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 8; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 3: Comparison: Changes in Home Diastolic Blood Pressure From Baseline; The null hypothesis was that the mean changes in home DBP from the baseline are equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Week 12; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 4: Comparison: Changes in Home Diastolic Blood Pressure From Baseline; The null hypothesis was that the mean changes in home DBP from the baseline are equal to 0; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — Last Day; A one-sided paired t-test was performed to test the hypothesis

ADVERSE EVENTS:
Description: The frequency of adverse events during the study.
Arm/Group | Amlodipine 10 mg Tablet
Serious Adverse Events (participants affected / at risk) | 78/13343
Other Adverse Events (participants affected / at risk) | 250/13343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine 10 mg Tablet (N=13343)
Enteritis infectious (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intracranial haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Marasmus (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 7 (7)
Epilepsy (Nervous system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 6 (6)
Loss of consciousness (Nervous system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Aphagia (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine 10 mg Tablet (N=13343)
Bronchitis (Infections and infestations) | 17 (17)
Diabetes mellitus (Metabolism and nutrition disorders) | 22 (22)
Headache (Nervous system disorders) | 14 (14)
Dizziness (Nervous system disorders) | 45 (45)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (15)
Constipation (Gastrointestinal disorders) | 16 (16)
Oedema (General disorders) | 14 (14)
Oedema peripheral (General disorders) | 85 (85)
Blood pressure decreased (Investigations) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.